CLINICAL TRIAL: NCT07084142
Title: Developing "A Digital Shared Decision-Making Aid to Improve Patient-Centered Outcomes in Implantable Cardioverter-Defibrillator (ICD) Decisions Among Older Patients"
Brief Title: Developing a Digital Aid to Improve ICD Decisions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of California, San Francisco (Other); East Carolina University (Other)
Responsible Party: Principal Investigator, Randall Stafford, Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB-79108; R01HL173578 (NIH)
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure and Reduced Ejection Fraction
Keywords: heart failure; HFrEF; sudden cardiac death; patient education; shared decision-making; arrhythmia; implantable cardioverter-defibrillator
MeSH Terms: conditions — Heart Failure, Systolic; Heart Failure; Death, Sudden, Cardiac; Arrhythmias, Cardiac | interventions — Amyloid; Defibrillators, Implantable

STUDY DESIGN:
Intervention Model Description: Three-arm randomized, parallel clinical trial. Arm A: digital decision-making tool with personalized risk information, Arm B: digital decision-making tool without personalized risk information, and Arm C: usual clinical care without digital tool use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Exposure to digital decision-making app with personal risk information (Experimental): The participant will use the pre-visit, participant-facing app with personal risk information derived from participant characteristics. During a clinical encounter, the clinician will have access to an abbreviated clinician-facing digital tool that displays the same personalized information.
  Interventions: Other: Online, patient-facing decision-making aid (app) with personalized risk information.; Device: Implantable Cardioverter Defibrillator (ICD)
- Use of a digital decision-making app without personalized risk information. (Experimental): The participant will use the pre-visit, participant-facing app without personal risk information. During a clinical encounter, the clinician will have access to an abbreviated clinician-facing digital tool.
  Interventions: Device: Implantable Cardioverter Defibrillator (ICD); Other: Online, patient-facing decision-making app without personalized risk information.
- Usual clinical care (Placebo Comparator): Participant will receive usual clinical care without use of the digital decision-making app.
  Interventions: Device: Implantable Cardioverter Defibrillator (ICD)

INTERVENTIONS:
Other: Online, patient-facing decision-making aid (app) with personalized risk information. — The online, patient-facing decision-making aid will have the following features:
  1. Clinical Data Input,
  2. Introduction via Animated Video,
  3. Common Questions,
  4. Check-In Quiz,
  5. Risk and Values Exploration based on patient specific information,
  6. Wrap-Up,
  7. Patient-Physician Worksheet,
  These steps will be completed by the patient in advance of a provider visit where a shared-decision making process will decide whether an ICD is an appropriate sudden cardiac death-prevention strategy to pursue.
  Arms: Exposure to digital decision-making app with personal risk information
Device: Implantable Cardioverter Defibrillator (ICD) — Some participants, in their course of medical care unrelated to the study intervention, will undergo implantation of an ICD.
Other: Online, patient-facing decision-making app without personalized risk information. — The online, patient-facing decision-making aid will have the following features: 1) Clinical Data Input, 2) Introduction via Animated Video, 3) Common Questions, 4) Check-In Quiz, 5) Generic Risk and Values Exploration without patient specific information, 6) Wrap-Up, 7) Patient-Physician Worksheet, These steps will be completed by the patient in advance of a provider visit where a shared-decision making process will decide whether an ICD is an appropriate sudden cardiac death-prevention strategy to pursue.
  Arms: Use of a digital decision-making app without personalized risk information.

SUMMARY:
Advanced heart failure, affecting 7 million Americans, has multiple causes and results in greatly increased risk of disability and death. A major problem is sudden cardiac death, when the damaged heart develops an abnormal pattern of electrical conduction that can result in cessation of heart activity. While placement of an Implantable Cardioverter-Defibrillator (ICD) in a patient's chest can help prevent sudden cardiac death, these devices have several important downsides. This protocol focuses on development of a digital decision aid that helps heart failure patients make informed decisions that balance the benefits and downsides of ICD placement. This protocol covers the use of participant surveys, focus groups, and interviews to obtain the needed background information to guide the development of this digital tool, which will be subsequently tested against usual care in a randomized clinical trial. The study design is best described as a mixed methods evaluation and refinement of a digital app to improve ICD decision-making. In the future, the present protocol will be modified to create a new protocol that covers the needed human subjects requirements for performance of this clinical trial.

DETAILED DESCRIPTION:
Advanced heart failure, affecting 7 million Americans, has multiple causes and results in greatly increased risk of disability and death. A major problem is sudden cardiac death, when the damaged heart develops an abnormal pattern of electrical conduction that can result in cessation of heart activity. While placement of an Implantable Cardioverter-Defibrillator (ICD) in a patient's chest can help prevent sudden cardiac death, these devices have several important downsides. This protocol focuses on development of a digital decision aid that helps heart failure patients make informed decisions that balance the benefits and downsides of ICD placement. This protocol covers the use of participant surveys, focus groups, and interviews to obtain the needed background information to guide the development of this digital tool, which will be subsequently tested against usual care in a randomized clinical trial. In the future, the present protocol will be modified to create a new protocol that covers the needed human subjects requirements for performance of this clinical trial.

Participants with heart failure who agree to participate will be recorded in a REDCap system database. The investigators will document in a recruitment tracking log all potentially eligible participants found to be ineligible or who decline participation. The reason for ineligibility or reason for decline will be captured along with age, gender, and race/ethnicity. At the time of their enrollment, the investigators will collect additional information from each participant about their employment status (full-time or part-time employment, no employment, retired), education (no postsecondary education, some postsecondary education), household size (living alone, living with at least one other person).

Participants with heart failure will be asked if they are willing to be interviewed, participate in focus groups, or complete surveys to determine their views on 1) which elements of patient outcome questionnaires are important to them; 2) which decision aid components or educational tools they like or find valuable. Interactions with participants will include open-ended interviews, focus groups, and surveys. These interviews, focus groups, and surveys will be conducted by study staff to help develop a patient-centric shared decision making software tool. Development will occur iteratively with new testing after any modifications. The same individuals may be asked to re-test the app following alterations.

Collaborating teams from UC San Francisco (Site PI: Daniel Morin, MD, MPH) and East Carolina University (Site PI: Samuel Sears, PhD) will join the study before the third month of operation. The participation of these clinical sites is not needed in the first steps on digital tool development. By successfully initiating the project at Stanford, the process of initiation at the clinical sites will be facilitated and is consistent with the mandated use of a single IRB for the three sites.

ELIGIBILITY:
Developmental Testing will attempt to abide by eligibility criteria identical to the planned criteria for the subsequent RCT, but may strategically deviate from these criteria to enhance the testing and development process.

Inclusion Criteria:

* Meets or approximates minimal criteria for primary prevention ICD placement. ● Left Ventricular Ejection Fraction (LVEF) <35%.
* Clinical diagnosis of Heart Failure:
* Patients with severe ischemic dilated cardiomyopathy and underlying NYHA
* Class II or III Heart Failure, OR, Patients with severe nonischemic dilated cardiomyopathy and underlying NYHA Class II or III Heart Failure.
* Age ≥ 70 years old.
* Able to consent in English, Mandarin or Spanish and follow study instructions.

Exclusion Criteria:

The exclusion criteria include any of the following:

* Past ICD implantation (not including pacemakers).
* Any indication for secondary prevention of SCD via ICD implantation.
* History of mechanical valve replacement.
* History of recent myocardial infarction within the last 40 days.
* History of recent revascularization within the past 90 days.
* History of familial or genetic disorders with a high-risk of ventricular arrhythmias, such as the long QT syndrome (LQTS) or hypertrophic cardiomyopathy (HCM).
* Any factors contraindicating ICD placement.
* Less than 6 months life expectancy and other clinical consideration,
* Unwilling or unable to consider ICD,
* Any contraindications to ambulati

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Decisional Conflict Scale (DCS) | Immediately after decision-making visit as well as at 3 months.
  The Decisional Conflict Scale is a validated, 16-item questionnaire scale assessing whether a participant feels conflicted regarding a past medical decision. The range is 0 to 100 with higher scores indicating more conflict, a negative outcome.

OTHER OUTCOMES:
System Usability Scale (SUS) | Day 1 (SUS will be assessed immediately following testing of the app, or a specific module of the app)
  System Usability Scale (SAS) Standard Version is a metric for determining the ease of use of an online app. The app development process will focus on optimizing the user experience in each module of the proposed application. With a range of 0 to 100, a higher score is better. A score above 70 is considered acceptable.

CONTACTS AND LOCATIONS:
Overall Officials: Randall S Stafford, MD, PhD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - Eastern Carolina University, Greenville, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request after January 1, 2027, IPD will be provided without cost.
Supporting Information: Study Protocol
Time Frame: IPD from this developmental stage will be available after January 1, 2027 for a period of at least 5 years.
Access Criteria: Electronic access will be provided to IPD upon approval of reasonable requests.

DOCUMENTS (2):
  • Informed Consent Form: Part 1 (2025-07-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT07084142/ICF_000.pdf
  • Informed Consent Form: Part 2 (2025-07-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT07084142/ICF_001.pdf